CLINICAL TRIAL: NCT06974253
Title: Morphological Characteristics of Anterior Maxillary Anchorage Sites and Application of Dynamic Navigation in Full-Arch Dental Implant Placement
Brief Title: Morphological Characteristics of Anterior Maxillary Bone and Dynamic Navigation in Full-Arch Implant Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Bui Tan Lam, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25213-DHYD
Record Dates: First submitted 2025-04-30; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Atrophy of Edentulous Maxillary Alveolar Ridge; Alveolar Bone Atrophy
Keywords: Nasopalatine Implant; Trans-sinus Implant; Trans-nasal Implant; Piriform Rim Implant
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Full-arch dental implant treatment with dynamic navigation (Experimental): This study involves placing three types of implants-nasopalatine, trans-sinus, and trans-nasal implants-using dynamic navigation in patients with complete maxillary edentulism and severe bone resorption. The primary goal is to assess the accuracy of implant placement and the clinical effectiveness of these implants for full-arch rehabilitation. Key measurements, such as 3D deviation, lateral and vertical linear deviation, and angular deviation, will be analyzed to compare the actual and planned implant positions. This study aims to evaluate the precision and success of dynamic navigation-assisted implant placement in patients with significant bone loss.
  Interventions: Procedure: Nasopalatine Implants, Trans-Sinus Implants, and Trans-Nasal Implants for Full-Arch Rehabilitation

INTERVENTIONS:
Procedure: Nasopalatine Implants, Trans-Sinus Implants, and Trans-Nasal Implants for Full-Arch Rehabilitation — Pre-surgery (Implant Placement):
  Clinical examination, panoramic radiography, film guide creation, and CBCT imaging will be performed. Based on CBCT data and the film guide, bone measurements will be taken, and a treatment plan with virtual implants will be developed. 4-6 pilot holes will be made, adjusting for critical structures like the maxillary sinus, inferior alveolar nerve, and planned implant sites. Full blood count and coagulation tests will be done.
  During Surgery:
  Implant surgery will be performed under local anesthesia/sedation. Incision and mucosal flap reflection will expose the implant site. A clip will be fixed to the anterior maxilla with screws, connected to the monitoring device. The dynamic navigation system will guide the placement of nasopalatine, trans-sinus, and trans-nasal implants, ensuring optimal placement.
  Post-surgery:
  Post-operative CBCT will be performed to check the implant positions, confirming the accuracy of the implant placement.

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of dynamic navigation in full-arch dental implant placement in patients with complete maxillary edentulism. The main questions it aims to answer are:

* the accuracy of nasopalatine implants, trans-sinus implants, and trans-nasal implants placement in the anterior maxillary bone with dynamic navigation
* the clinical effectiveness of nasopalatine implants, trans-sinus implants, and trans-nasal implants in full-arch rehabilitation
* the correlation between the anatomical features of the nasal cavity and the anterior sinus wall on CBCT images and their influence on nasopalatine implants, trans-sinus implants, and trans-nasal implants position

DETAILED DESCRIPTION:
This study aims to explore the anatomical features of the anterior maxillary bone and then apply dynamic navigation technology for full-arch dental implant placement. The primary goal is to assess how dynamic navigation can improve the precision and success of implant placement in patients with complete edentulism or significant bone resorption in the upper jaw.

1. Objectives:

   * To analyze the anatomical features of the nasopalatine canal and the anterior sinus wall using CBCT imaging to guide full-arch implant placement.
   * To evaluate the accuracy of implant surgeries, including the placement of nasopalatine implants, trans-sinus implants, and trans-nasal implants, with the assistance of dynamic navigation systems.
   * To assess the clinical effectiveness of nasopalatine implants, trans-sinus implants, and trans-nasal implants in full-arch rehabilitation.
   * To investigate the correlation between the anatomical features of the nasal cavity and the anterior sinus wall on CBCT images and their influence on implant placement outcomes.
2. Clinical Study:

Study Type: Clinical Trials Study. Study Period: From 2024 to 2027.

Study Locations:

* The Center of Dentistry, University of Medicine and Pharmacy at Ho Chi Minh City
* Van Hanh General Hospital Sampling Method: Convenience sampling.

Study Subjects:

The study will involve a convenience sample of patients with complete or partial edentulism, who require tooth extraction and full-arch rehabilitation with implants. These patients will receive treatment at the Center of Dentistry, University of Medicine and Pharmacy at Ho Chi Minh City, and Van Hanh General Hospital from May 2025 to December 2027. Each patient may have multiple study units (implants) depending on the treatment plan.

Inclusion Criteria:

* Patients aged 18 years and above.
* Good overall health (Class 1 and 2 according to the American Society of Anesthesiologists classification system).
* Patients with complete edentulism of the upper jaw, classified as Class IV to VI according to Cawood and Howell.

Exclusion Criteria:

* Systemic or local conditions that may interfere with surgery, healing, or bone integration, such as cardiovascular diseases, diabetes, bone-related diseases, or medications affecting bone metabolism.
* Patients who smoke more than 10 cigarettes per day or have untreated acute infections at the planned implant site.
* Patients with a mouth opening limited to less than 40mm.

Study Procedure:

Pre-surgery (Implant Placement):

* Clinical examination, panoramic radiography, fabrication of a film guide, and CBCT imaging with the film guide will be performed.
* Based on CBCT data and the film guide, bone measurements will be taken, and a treatment plan will be created using virtual implants with appropriate positions and sizes.
* 4-6 pilot holes will be placed for implant placement, adjusted to avoid critical anatomical structures like the maxillary sinus and inferior alveolar nerve.
* Full blood count and coagulation tests will be conducted.

During Surgery:

* Implant surgery will be performed under local anesthesia or sedation.
* An incision and full mucosal flap reflection will expose the implant site.
* A clip will be secured to the anterior bone region of the maxilla using at least two screws. The clip will be connected to the handle and the patient monitoring device, which will be attached to the surgical drill.
* The dynamic navigation system tool will be adjusted, and the synchronization of the system's landmarks will be performed.
* Drilling and implant placement will be guided using the dynamic navigation system.
* The primary stability of the implants will be measured. Depending on the stability, the implants will be connected to either a healing cap or multi-unit abutment.
* Suturing will be performed.

Post-surgery:

* Post-operative CBCT imaging will be performed.
* Post-operative care will include prescribed medications, cold compresses for the first day, and warm compresses starting from the second day after surgery. Gentle cleaning of the surgical site will be advised. Provisional restorations will be provided.
* Follow-up visits will be scheduled on the 3rd, 7th, 14th, 1st month, 3rd month, and 6th month after surgery. Permanent restoration will be performed on the implants at the 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Good overall health (Class 1 and 2 according to the American Society of Anesthesiologists classification system)
* Clinical diagnosis of complete edentulism of the upper arch classified as Class IV to VI according to Cawood and Howell

Exclusion Criteria:

* Systemic or local conditions that may affect surgery, wound healing, or bone integration, such as cardiovascular diseases, diabetes, bone-related diseases, or medication affecting bone metabolism
* Smoking more than 10 cigarettes per day
* Presence of acute infections in the planned implant site
* Limited mouth opening of less than 40mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Bone-to-implant contact | From enrollment to the end of surgery (second CBCT)
  Radiographs are analyzed to measure the bone level around the implant (mm). Bone-to-implant contact (BIC) is a crucial parameter used to evaluate the success and stability of dental implants.
3D Deviation at Apex | From enrollment to the end of surgery (second CBCT)
  This measures the 3D deviation at the apex (bottom) of the implant site, which similarly involves assessing the horizontal and vertical position, along with depth, between the planned and actual implant positions at the tip of the implant (mm).
3D Deviation at Coronal | From enrollment to the end of surgery (second CBCT)
  This measures the three-dimensional (3D) deviation between the planned implant position and the actual implant position at the coronal (top) aspect of the implant site (mm). It involves assessing discrepancies in the X, Y, and Z axes (horizontal, vertical, and depth).
Lateral Linear Deviation | From enrollment to the end of surgery (second CBCT)
  This measures the horizontal distance (in the X or Y axis) between the planned implant position and the actual position (mm), specifically at the coronal or apical levels, and refers to any shift in the lateral direction.
Vertical Linear Deviation | From enrollment to the end of surgery (second CBCT)
  This measures the vertical distance between the planned and actual positions of the implant, assessing any deviation in the upward or downward direction along the Z axis (mm).
Angular Deviation | From enrollment to the end of surgery (second CBCT)
  This measures the angular (°) difference between the planned angle of the implant and the actual angle of the implant at the coronal or apical level. It helps assess how well the implant's rotation and orientation match the planned design.

SECONDARY OUTCOMES:
Implant Survival Rate at 6 months post-surgeryy | From enrollment to the prosthetic stage (6 months post-surgery)
  Implant survival rate refers to the proportion of implants that remain in place without failure throughout the study period. An implant is considered to have survived if it remains functional, does not exhibit signs of failure (such as infection or implant loosening), and is not removed due to complications. The survival rate is typically measured as a percentage of implants that remain in place compared to the total number of implants placed. This measure provides a basic indication of the long-term effectiveness of the implant procedure.
Stability of Implant | From enrollment to the prosthetic stage (6 months post-surgery)
  Implant stability refers to the degree of primary and secondary integration between the implant and surrounding bone. This is evaluated using measures such as resonance frequency analysis during placement (ISQ). Primary stability occurs immediately after placement, while secondary stability refers to the osseointegration process during healing.
Torque value | In the surgery
  This is evaluated using measures of torque (Ncm) values during placement.

CONTACTS AND LOCATIONS:
Overall Officials: Lam Tan Bui, MSc, Principal Investigator — Faculty of Dentistry, University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- Faculty of Dentistry, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
We intend to share IPD regarding the deviation in implant positioning from planned data. No personally identifiable information (PII) will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: May 2025 - February 2028
Access Criteria: The IPD and supporting information will be accessible to researchers, regulatory bodies, and other authorized individuals involved in the study. Access will be granted to those who have received approval from the ethics committee or relevant regulatory authorities. These individuals will be able to access the data via a secure, password-protected portal or system provided by the study team. All users will be required to sign a data sharing agreement to ensure confidentiality and compliance with the relevant data protection regulations.

REFERENCES:
- [Background] Nunes M, de Araujo Nobre M, Camargo V. All-on-4 Hybrid with Extra-Long Transnasal Implants: Descriptions of the Technique and Short-Term Outcomes in Three Cases. J Clin Med. 2024 Jun 6;13(11):3348. doi: 10.3390/jcm13113348. PMID 38893060
- [Background] Almeida PHT, Cacciacane SH, Arcazas Junior A. Extra-long transnasal implants as alternative for Quad Zygoma: Case report. Ann Med Surg (Lond). 2021 Jul 27;68:102635. doi: 10.1016/j.amsu.2021.102635. eCollection 2021 Aug. PMID 34386227
- [Background] Singhal MK, Dandriyal R, Aggarwal A, Agarwal A, Yadav S, Baranwal P. Implant Placement into the Nasopalatine Foramen: Considerations from Anatomical and Surgical Point of View. Ann Maxillofac Surg. 2018 Jul-Dec;8(2):347-351. doi: 10.4103/ams.ams_161_17. PMID 30693262
- [Background] Jensen OT, Cottam J, Ringeman J, Adams M. Trans-sinus dental implants, bone morphogenetic protein 2, and immediate function for all-on-4 treatment of severe maxillary atrophy. J Oral Maxillofac Surg. 2012 Jan;70(1):141-8. doi: 10.1016/j.joms.2011.03.045. Epub 2011 Jul 28. PMID 21802186
- [Background] Pena-Cardelles JF, Markovic J, De Souza A, Hamilton A, Lanis A, Gallucci GO. Survival, Success, and Neuropathic Alterations Related to Implant Placement Procedures in the Nasopalatine Canal: A Systematic Review and Meta-analysis. Int J Periodontics Restorative Dent. 2025 Nov 7;45(6):805-811. doi: 10.11607/prd.7168. PMID 39270594
- [Background] Nicoli G, Piva S, Ferraris P, Nicoli F, Jensen OT. Extra-Long Nasal Wall-Directed Dental Implants for Maxillary Complete Arch Immediate Function: A Pilot Study. Oral Maxillofac Surg Clin North Am. 2019 May;31(2):349-356. doi: 10.1016/j.coms.2019.01.004. PMID 30947851
- [Background] Malo P, Nobre Md, Lopes A. Immediate loading of 'All-on-4' maxillary prostheses using trans-sinus tilted implants without sinus bone grafting: a retrospective study reporting the 3-year outcome. Eur J Oral Implantol. 2013 Autumn;6(3):273-83. PMID 24179981
- [Background] Grandi T, Faustini F, Casotto F, Samarani R, Svezia L, Radano P. Immediate fixed rehabilitation of severe maxillary atrophies using trans-sinus tilted implants with or without sinus bone grafting: One-year results from a randomised controlled trial. Int J Oral Implantol (Berl). 2019;12(2):141-152. PMID 31090746